CLINICAL TRIAL: NCT04307706
Title: Effect of Interventions Based on Acceptance and Commitment Therapy Administered to Parents of Special Needs Children on Their Levels of Psychological Resilience, Depression, Anxiety, Stress and Caregiver Burden: A Randomised Controlled Trial
Brief Title: Using Acceptance and Commitment Therapy for Parents of Disabled Child
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ecem CICEK GUMUS, Research Assistant, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDK-2019-4588
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Acceptance and Commitment Therapy; Anxiety Depression; Caregiver Burden; Public Health Nurse; Stress; Special Needs Children; Caregiver Burnout
MeSH Terms: conditions — Caregiver Burden | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): ''Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Control group (No Intervention): Only data collection was carried out. No attempt was made by the researcher during the study.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group in six sessions. The duration of each session lasted on average 60-90 minutes. A session was held for each parent once a week.
  Arms: Intervention group

SUMMARY:
This study was carried out to determine the effect of ACT-based interventions applied to parents of special needs children (CSN) on their levels of psychological inflexibility, psychological resilience, depression, anxiety, stress, and caregiver burden.

DETAILED DESCRIPTION:
This research is a pretest, posttest, follow-up, randomized controlled experimental study. The research was carried out in Şehitkamil and Şahinbey districts, which are two central districts of Gaziantep Province. 60 parents with disabled children were included in the study (intervention: 30 parents, control: 30 parents). The research data was collected as pretest, posttest and follow-up test from the intervention group between April and December 2019, and the control group between April and September 2019 in three stages. Parental Identification Form, Acceptance and Action Questionnaire (AAQ-II), Depression, Anxiety and Stress Scale (DASS-21), Adult Psychological Resilience Scale (RSA-21) were used as data collection form. After the pre-test data was collected, the Acceptance and Commitment Therapy Based Intervention Program was applied to the intervention group in six sessions. The duration of each session lasted on average 60-90 minutes. A session was held for each parent once a week. The control group participated in the training carried out by the guidance service.

The intervention programme based on ACT was prepared with the aim of reducing levels of psychological inflexibility, caregiver burden, depression, anxiety and stress, and of increasing levels of psychological resilience in parents of CSN.

In the preparation of the interventions and planning of the sessions based on ACT, the researcher utilised studies in the literature and the basic ACT training she had received. After preparation of the ACT intervention protocol, it was given its final shape by obtaining the views of specialists working in this field. The sessions were prepared based on six components of psychological flexibility found at the basis of ACT.

Keywords: Acceptance and commitment therapy (ACT), special needs child, psychological inflexibility, resilience, depression-anxiety-stress levels, caregiver burden, public health nurse.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children at the Gaziantep Private Education Practice Schools I. and II. stage (the mother or father will be the person who is primarily responsible for the child's care).
* Those living in the central districts of Gaziantep province,
* Those who have not received any such training (ACT) or received any psychiatric treatment/support or therapy,
* There is currently no ongoing psychological or psychiatric treatment,
* Does not have problems such as substance/alcohol addiction,
* Without communication disabilities (hearing and speaking),
* Speaking Turkish,
* Literate,
* Parents who agreed to participate in the research

Exclusion Criteria:

* Parents with cognitive impairment (mental retardation or a psychiatric diagnosis),
* Parents who have previously received psychiatric support or therapy,
* Parents with problems such as substance/alcohol abuse,
* Has a communication disability (hearing-speaking),
* Using a language other than Turkish,
* Illiterate parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire (AAQ-II) | 8 months
  The Acceptance and Action Questionnaire consists of 7 items and evaluates information about psychological consistency. the minimum and maximum values of scale changes between 7 and 49 points. Interpretation of score for scale; the high total score obtained from the scale shows that the level of "psychological consistency" is also high.
Depression, Anxiety and Stress Scale (DASS-21) | 8 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Adult Psychological Resilience Scale (RSA-21) | 8 months
  The Adult Psychological Resilience Scale consists of 21 items and evaluates information about psychological resilience. Minimum 21 points and maximum 105 points are obtained from the scale. The high total score obtained from the scale indicates that the level of "psychological resilience" is high.
The Zarit Burden Scale | 9 months
  The Zarit Burden Interview consists of 22 items and evaluates information about caregiver burden.Interpretation of Score: 0 - 21 little or no burden, 21 - 40 mild to moderate burden, 41 - 60 moderate to severe burden, 61 - 88 severe burden. The higher the score obtained, the higher the burden level

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, University Boulevard, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04307706/Prot_000.pdf